CLINICAL TRIAL: NCT00187902
Title: Evaluation of NAATs for Detection of C. Trachomatis and N. Gonorrhoeae From Pharynx, Rectum, Glans & Urethra of MSM
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Julius Schachter, PhD, Univ of CA, San Francisco
Other Study IDs: H1079-26791-01
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Sexually Transmitted Diseases; Chlamydia; Gonorrhea
Keywords: Sexually Transmitted Diseases; Chlamydia trachomatis; Neisseria gonorrhoeae
MeSH Terms: conditions — Sexually Transmitted Diseases; Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — self-collected glans swab; clinician-collected rectal and pharyngeal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
Julius Schachter, PhD, from the Department of Laboratory Medicine at UCSF, and Jeffrey Klausner, MD, from the Department of Public Health, are conducting a study to evaluate a type of test (nucleic acid amplification test) for the detection of two sexually transmitted diseases, Chlamydia trachomatis and Neisseria gonorrhoeae, in men who have sex with men (MSM), using urine samples and swabs taken from the throat (pharynx), tip of penis (glans), and rectum. The use of nucleic acid amplification tests on these swabs is experimental, which means that the use of the tests for this purpose have not been approved by the Food & Drug Administration.

DETAILED DESCRIPTION:
For all subjects enrolled in the study, the following clinical data information will be obtained: 1) reason for exam, 2) subject's signs and symptoms and 3) clinical assessment.

For each subject enrolled in the study, three clinician-collected pharyngeal, four rectal swabs (three clinician-collected, 1 self-collected) specimens, one glans swab (self-collected) and a first catch urine specimen (approximately 25 ml) will be obtained. The collection order of the clinician collected swabs will be randomized.

Three pharyngeal swabs will be tested for: 1) CT/NG NAAT (TMA) at DPH, 2) NG culture at DPH and 3) NAATs for CT/NG (TMA, SDA) and CT culture at UCSF. Four rectal swabs will be tested for: 1) CT/NG NAAT (TMA) at DPH, 2) NG culture at DPH and 3) NAATs for CT/NG on Clinician- and self-collected rectal swab (TMA, SDA) and CT culture at UCSF. Self-collected glans swab and the FCU will be tested by NAATs for CT/NG (TMA, SDA) at UCSF. All NAAT specimens collected in a universal NAAT transport medium. After specimen processing, samples will be frozen at -70 C for discrepant analysis.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be a man who has sex with men (MSM). Subjects must provide verbal consent, must be able to submit all required specimens and must not have urinated within 1 hr prior to providing a study urine specimen.

Exclusion Criteria:

* Subjects are excluded if they do not have sex with men, refuse to give verbal consent, are unable to provide all required specimens and minimum specimen volume, have been on antibiotic therapy within the last 21 days, have urinated within 1 hr prior to submitting study specimens, and have already been evaluated as part of this trial. Subjects will be excluded if specimens are mishandled or inappropriately stored.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men who have sex with men (MSM) voluntarily presenting at the City STD clinic.
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2005-10; Primary Completion 2007-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Positive nucleic acid amplification result for Chlamydia trachomatis or Neisseria gonorrhoeae. | At enrollment/screening

CONTACTS AND LOCATIONS:
Overall Officials: Julius Schachter, PhD, Principal Investigator — University of California, San Francisco; Jeffrey D Klausner, MD, MPH, Principal Investigator — Department of Public Health, San Francisco, CA USA
Locations (1):
- City Clinic, San Francisco, California, United States

REFERENCES:
- [Background] Johnson RE, Newhall WJ, Papp JR, Knapp JS, Black CM, Gift TL, Steece R, Markowitz LE, Devine OJ, Walsh CM, Wang S, Gunter DC, Irwin KL, DeLisle S, Berman SM. Screening tests to detect Chlamydia trachomatis and Neisseria gonorrhoeae infections--2002. MMWR Recomm Rep. 2002 Oct 18;51(RR-15):1-38; quiz CE1-4. PMID 12418541
- [Background] Sexually transmitted diseases treatment guidelines 2002. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 May 10;51(RR-6):1-78. PMID 12184549
- [Background] Page-Shafer K, Graves A, Kent C, Balls JE, Zapitz VM, Klausner JD. Increased sensitivity of DNA amplification testing for the detection of pharyngeal gonorrhea in men who have sex with men. Clin Infect Dis. 2002 Jan 15;34(2):173-6. doi: 10.1086/338236. Epub 2001 Dec 7. PMID 11740704
- [Background] Van Der Pol B, Ferrero DV, Buck-Barrington L, Hook E 3rd, Lenderman C, Quinn T, Gaydos CA, Lovchik J, Schachter J, Moncada J, Hall G, Tuohy MJ, Jones RB. Multicenter evaluation of the BDProbeTec ET System for detection of Chlamydia trachomatis and Neisseria gonorrhoeae in urine specimens, female endocervical swabs, and male urethral swabs. J Clin Microbiol. 2001 Mar;39(3):1008-16. doi: 10.1128/JCM.39.3.1008-1016.2001. PMID 11230419
- [Background] Ciemins EL, Flood J, Kent CK, Shaw H, Rowniak S, Moncada J, Klausner JD, Schachter J. Reexamining the prevalence of Chlamydia trachomatis infection among gay men with urethritis: implications for STD policy and HIV prevention activities. Sex Transm Dis. 2000 May;27(5):249-51. doi: 10.1097/00007435-200005000-00002. PMID 10821595
- [Background] Centers for Disease Control and Prevention (CDC). High prevalence of chlamydial and gonococcal infection in women entering jails and juvenile detention centers--Chicago, Birmingham, and San Francisco, 1998. MMWR Morb Mortal Wkly Rep. 1999 Sep 17;48(36):793-6. PMID 10499782
- [Background] Moncada J, Chernesky M, McCormack W, Schachter J. Evaluation of the Gen-Probe Amplified Chlamydia trachomatis Assay on self-collected vaginal swabs from asymptomatic young females. In: Stephens RS, Byrne GI, Christiansen G, Clarke IN, Grayston JT, Rank RG, et al., editors. Chlamydial Infections: Proceedings of the Ninth International Symposium on Human Chlamydial Infection. San Francisco: International Chlamydia Symposium, 1998:595-8.
- [Background] Ostergaard L, Agner T, Krarup E, Johansen UB, Weismann K, Gutschik E. PCR for detection of Chlamydia trachomatis in endocervical, urethral, rectal, and pharyngeal swab samples obtained from patients attending an STD clinic. Genitourin Med. 1997 Dec;73(6):493-7. doi: 10.1136/sti.73.6.493. PMID 9582468
- [Background] Schachter J. DFA, EIA, PCR, LCR and other technologies: what tests should be used for diagnosis of chlamydia infections? Immunol Invest. 1997 Jan-Feb;26(1-2):157-61. doi: 10.3109/08820139709048923. PMID 9037620
- [Background] Rompalo AM, Price CB, Roberts PL, Stamm WE. Potential value of rectal-screening cultures for Chlamydia trachomatis in homosexual men. J Infect Dis. 1986 May;153(5):888-92. doi: 10.1093/infdis/153.5.888. PMID 3084665